CLINICAL TRIAL: NCT04790409
Title: Department of Medical Oncology, Zhejiang Cancer Hospital
Brief Title: Sintilimab Combined With Anlotinib in Advanced NSCLC With EGFR Uncommon Mutations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Fan Yun, MD, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2019-81
Record Dates: First submitted 2021-02-18; First posted 2021-03-10 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — sintilimab; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab with anlotinib (Experimental): Patients received sintilimab (anti-PD-1) combined with anlotinib (multi-target anti-angiogenesis).
  Interventions: Drug: sintilimab and anlotinib

INTERVENTIONS:
Drug: sintilimab and anlotinib — This study was a one-arm, open-label, phase II study of PD-1 monoclonal antibody combined with ilotinib in the treatment of advanced EGFR rare-mutant non-small cell lung cancer (NSCLC). 21 patients enrolled in the study who underwent platinum-containing systemic chemotherapy and EGFR-TKI failure were enrolled in the study.

SUMMARY:
This study was a single-arm, open-label, phase II study of PD-1 monoclonal antibody combined with anlotinib in the treatment of advanced non-small cell lung cancer (NSCLC) with EGFR uncommon mutations. Twenty-one patients of NSCLC harboring rare EGFR mutations after previous treatments, including a platinum-based regimen and a targeted treatment (regardless of EGFR Ex20ins), were enrolled. Patients received sintilimab (anti-PD-1) combined with anlotinib (multi-target anti-angiogenesis). The primary endpoint was the objective response rate (ORR) based on RECIST 1.1. Secondary goals included progression-free survival (PFS), overall survival (OS), disease control rate (DCR) based on RECIST 1.1; safety Sex and tolerance. Exploratory objectives include the use of tumor tissue and plasma specimens to detect biomarkers predicting the efficacy of sidilimumab: including but not limited to tumor mutation burden (TMB), PD-L1 expression, etc.; exploring potential predictions in peripheral blood. Biomarkers for anti-group efficacy, including but not limited to TCR.

DETAILED DESCRIPTION:
This clinical trial (NCT04790409) entitled " Sintilimab Combined with Anlotinib in Advanced NSCLC with EGFR Uncommon Mutations" has been approved by the Ethics Committee of Zhejiang Cancer Hospital in June 12, 2019 (IRB-2019-81). Meanwhile, we registered our project information on the ClinicalTrials.gov PRS in June, 2019 and obtained the status of "approved". In this study, the first patient received treatment on August 26, 2019. However, due to inexperience and misunderstanding, we wrongly missed the next stage of "released" in PRS. Until we realize our mistakes, the initial release time can only be on 02/18/2021. Therefore, we amend the initial release time here.

ELIGIBILITY:
Inclusion Criteria:

1. Sign written informed consent before any trial-related processes are implemented;
2. Age ≥ 18 years old and ≤ 75 years old;
3. Life expectancy exceeds 3 months;
4. The investigator confirmed at least one measurable lesion according to the RECIST 1.1 standard. A measurable lesion located in the field of previous radiation therapy or after local treatment may be selected as a target lesion if it is confirmed to have progressed;
5. Patients with treated metastatic or recurrent (stage IV) NSCLC confirmed by histology or cytology according to the International Association for the Study of Lung Cancer and the American Association for the Classification of Cancer Classification, 8th edition;
6. The Eastern Cancer Cooperative Group (ECOG) has a fitness status score of 0 or 1;
7. Patients with genetic testing (allowing PCR and NGS detection methods) confirmed uncommon mutations (EGFR G719X, L861Q, S768I, and 20ins et al.), patients can accept two or more types of EGFR rare co-mutation. Populations with the primary EGFR T790M mutation can also be included in the study.
8. Patients who have experienced disease progression after at least two treatment regimens for advanced/metastatic disease must include a platinum-containing systemic chemotherapy and an EGFR-TKI treatment. Patients with EGFR 20ins who have experienced disease progression only after platinum-containing systemic chemotherapy.
9. Hematological function is sufficient, defined as absolute neutrophil count ≥1.5×109 /L, platelet count ≥100 ×109 /L, hemoglobin ≥90g/L (no history of blood transfusion within 7 days);
10. Hepatic function is adequate, defined as all patients with total bilirubin levels ≤ 1.5 times normal upper limit (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN, or for patients with liver metastases , AST and ALT levels ≤ 5 times ULN;
11. adequate renal function, defined as creatinine clearance ≥ 45 ml/min (Cockcroft-Gault formula);
12. Coagulation function is adequate, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; if the subject is receiving anticoagulant therapy, as long as the INR or PT is within the range of anticoagulant drugs can;
13. Female subjects of childbearing age should be negative for urine or serum pregnancy test within 3 days prior to receiving the first study drug. If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is required;
14. If there is a risk of conception, male and female patients need to use high-efficiency contraception (ie, an annual failure rate of less than 1%) and continue until at least 180 days after stopping the trial treatment; Note: If abstinence is normal for the subject Lifestyle and preferred methods of contraception can be used as a method of contraception.

Exclusion Criteria:

1. Histology is NSCLC, if there are small cell carcinoma, neuroendocrine carcinoma, sarcoma components, it can not be included;
2. Patients with known EGFR-sensitive mutations (19-Del and L858R);
3. Cavity lung squamous cell carcinoma, or non-small cell lung cancer patients with hemoptysis (>50 mL/day);
4. Patients whose tumor has invaded an important blood vessel or who is judged by the investigator to have major bleeding during the follow-up study;
5. Patients with any signs or history of bleeding physique;
6. Currently participating in interventional clinical research treatment, or receiving other research drugs or research equipment within 4 weeks prior to the first dose;
7. Previously received the following treatments: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or against another stimulus or synergistic inhibition of T cell receptors (eg CTLA-4, OX-40, CD137) drug;
8. Received a proprietary Chinese medicine or immunomodulatory drug (thymosin, interferon, interleukin, etc.) with anti-cancer indications within 2 weeks before the first dose, or received major surgery within 3 weeks before the first dose;
9. Received a physical organ or blood system transplant;
10. There is clinically uncontrollable pleural effusion/peritoneal effusion (patients who do not need drainage or stop drainage and have no significant increase in 3 days of effusion can be enrolled);
11. The tumor compresses important organs (such as the esophagus) around it and is accompanied by related symptoms, oppression of the superior vena cava or invasion of the mediastinal vessels, heart, etc.;
12. Class III-IV congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmias;
13. Any arterial thrombosis, embolism or ischemia occurred within 6 months prior to enrollment, such as myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack. A history of deep vein thrombosis, pulmonary embolism, or any other severe thromboembolism within 3 months prior to enrollment (implanted IV port or catheter-derived thrombosis, or superficial vein thrombosis is not considered a "serious" thrombosis embolism);
14. It is known that there is an allergic reaction to the active ingredient of sindril mAb and or any excipients;
15. Active autoimmune diseases requiring systemic treatment (eg, using disease-modifying drugs, corticosteroids or immunosuppressants) within 2 years prior to the first dose. Alternative therapies (such as thyroxine, insulin, or physiological doses of corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatments;
16. Patients who require long-term systemic use of corticosteroids. Patients with intermittent use of bronchodilators, inhaled corticosteroids, or topical corticosteroids due to COPD or asthma may be enrolled.
17. has not fully recovered from toxicity and/or complications caused by any intervention prior to initiation of treatment (ie, ≤1 or baseline, excluding fatigue or alopecia);
18. diagnosis within 5 years prior to initial dosing For other malignancies, it does not include radical cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ. If more than 5 years before the drug is diagnosed as other malignant tumors or lung cancer, pathological or cytological diagnosis of recurrent metastatic lesions is required;
19. symptomatic central nervous system metastasis. For patients with asymptomatic brain metastases or brain metastases with stable symptoms after treatment, as long as all the following criteria are met, participate in this study: measurable lesions outside the central nervous system; no midbrain, pons, cerebellum, meninges, Medulla or spinal cord metastasis; maintain clinical stability for at least 2 weeks; stop hormone therapy 14 days before the first study drug;
20. One year before the first dose, a history of non-infectious pneumonia requiring corticosteroid treatment or the presence of non-infectious pneumonia;
21. active infections requiring treatment or systemic anti-infectives used within one week prior to first administration;
22. There are known cases of mental illness or substance abuse that may have an impact on compliance with the test requirements;
23. A history of human immunodeficiency virus (HIV) infection (ie, HIV 1/2 antibody positive), known syphilis infection (positive syphilis antibody), and active tuberculosis are known.
24. Untreated active hepatitis B; Note: Hepatitis B subjects meeting the following criteria are also eligible for inclusion:

    The HBV viral load must be <1000 copies/ml (200 IU/ml) or below the lower limit of detection before the first dose. Subjects should receive anti-HBV treatment during the entire study chemotherapy drug treatment to avoid viral reactivation. For subjects with anti-HBc(+), HBsAg(-), anti-HBs(-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but viral reactivation is closely monitored;
25. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
26. Vaccination with live vaccine within 30 days prior to first dose; Note: Injectable inactivated virus vaccine for seasonal influenza is permitted; however, live attenuated influenza vaccine for intranasal administration is not permitted;
27. There are medical history, disease, treatment, or laboratory abnormalities that may interfere with the test results, hinder the subject's full participation in the study, or the investigator believes that participating in the study is not in the best interest of the subject.
28. Local or systemic diseases caused by non-malignant tumors, or secondary reactions to cancer, and may lead to higher medical risks and/or uncertainty in survival assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | objective response rate (ORR) through study completion, an average of 1 year
  objective response rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Yun Fan, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen K, Xu Y, Huang Z, Yu X, Hong W, Li H, Xu X, Lu H, Xie F, Chen J, Xu Y, Fan Y. Sintilimab plus anlotinib as second- or third-line therapy in metastatic non-small cell lung cancer with uncommon epidermal growth factor receptor mutations: A prospective, single-arm, phase II trial. Cancer Med. 2023 Oct;12(19):19460-19470. doi: 10.1002/cam4.6548. Epub 2023 Sep 18. PMID 37723837